CLINICAL TRIAL: NCT06581900
Title: Study of Vitamin B12 Metabolism in Children With Sickle Cell Disease Exposed to MEOPA , a Prospective Study at Reims University Hospital
Brief Title: Study of Vitamin B12 Metabolism in Children With Sickle Cell Disease Exposed to MEOPA
Acronym: DREPAM
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA24081*
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cells Patients
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle cells patients exposed to MEOPA: Sickle cells patients exposed to MEOPA during an hospitalization for a CVO
  Interventions: Other: Vitamin B12

INTERVENTIONS:
Other: Vitamin B12 — Quantification of Vitamin B12

SUMMARY:
Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis (Limit : 5000 characters) The sickle cells anemia is a monogenic disease linked to the presence of Hemoglobin S due to a mutation in the Hemoglobin Beta chain. The lack of circulating oxygen induces a polymerization of the Hemoglobin S which change the red cell conformation into sickle. Those cells interact and causes vaso-occlusive crisis (CVO).

The MEOPA is a medical gas used as an antalgic and a sedative especially in sickle cells disease patients. The nitrous oxide, oxide the cobalt ion in the vitamin B12 which inactivate it irreversibly creating a functional deficiency.

During the metabolism of vitamin B12, homocysteine is transformed in methionine which is used in to form the myelin sheath and helped in producing DNA. Numerous studies already shown that the longer the exposition to MEOPA is the greater the functional deficiency of vitamin B12 occur.

A few studies shown a symptomatic deficiency of vitamin B12 due to the exposition of MEOPA in sickle cells patient but there is no explanation on the necessary amount of exposure or if some patients are more at risk. When there is a deficiency of vitamin B12 the symptoms can go from a simple orthostatic hypotension to a combined spinal sclerosis.

The participation to the study will be proposed to every patient hospitalized for a CVO in the follow up of the emergency room visit or directly in pediatric reanimation. During a usual blood test, a small amount of blood (4mL) will be collected in addition to dose the Vitamin B12, the vitamin B9, the homocysteine, and the methionine. A small amount of urine will also be collected to dose the methylmalonic acid, all those elements are a part of the metabolism of B12 vitamin.

The same sample will be taken on the day of departure of the hospital. During the hospitalization the pain management, a daily neurological exam, and the exposition to the MEOPA will be assessed meticulously.

An appointment will take place at 7 days and at one month after the hospital departure to evaluate the possible neurological defect.

Each patient can only be included once.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cells patient
* Age between 2 and 18 years old
* Being affiliated with social security

Exclusion Criteria:

* Having a neurological defect prior to the study
* Being against the collection of blood or data

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patient hospitalized for a CVO in the follow up of the emergency room visit or in pediatric reanimation
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who will present a Vitamin B12 deficiency | Day 15
  Limit : Vitamin B12 <191pg/mL or homocysteine > 10micromol/L in children under 15 years old or > 15 micromol/L for children over 15 years old.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided